CLINICAL TRIAL: NCT06841614
Title: Evaluation of the Efficacy of a Post-exposure Prophylaxis (PEP) Strategy in Contacts at High Risk of Developing Ebola Virus Disease (EVD)
Brief Title: EBOla Post-Exposure Prophylaxis
Acronym: EBO-PEP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Alliance for International Medical Action (Other); Centre de Recherche et de Formation en Infectiologie de Guinée (CERFIG) (Unknown); Medecins Sans Frontieres, Netherlands (Other); Barcelona Institute for Global Health (Other); University of Bordeaux (Other); INSERM UMR S 1136 (Other); Agence Nationale de Sécurité Sanitaire de Guinée (ANSS) (Unknown); National Institute for Biomedical Research DRC (Unknown); Cheikh Anta Diop University, Senegal (Other); PACCI Program (Other); The PANdemic preparedness plaTform for Health and Emerging infectious Response (Unknown); University of Sierra Leone College of Medicine and Allied Health Sciences (Unknown); National Public Health Institute of Liberia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 0515s EBO-PEP
Record Dates: First submitted 2025-01-28; First posted 2025-02-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Ebola Virus Disease
Keywords: Ebola Virus Disease; EBOV; High-Risk contact; Post-Exposure Prophylaxis
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — atoltivimab, maftivimab, and odesivimab-ebgn drug combination

STUDY DESIGN:
Intervention Model Description: The total follow-up duration for trial participants is 60 days. All participants are followed daily for a minimum of 21 days.
  Some visits are conducted in person at the investigation site, also called the Post-Exposure Prophylaxis (PEP) center:
  * at Day 5, Day 10, and Day 21 for the ERV arm,
  * at Day 5, Day 10, Day 21, and Day 56 for the ERV+IMZ arm. Other visits are conducted at home or by phone, in collaboration with the Ministry of Health's surveillance team.
  Participants in the ERV+IMZ arm have an in-person visit at Day 56 to be revaccinated with the Ervebo vaccine to compensate for potential inhibition of the vaccine response when Ervebo is administered simultaneously with Inmazeb.
  Participants in the ERV arm have a phone visit at Day 56. For all participants, a phone visit is scheduled at Day 60. It corresponds to the last visit for all trial participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ervebo vaccine alone (Active Comparator): Administration of Ervebo vaccine (72 million PFU IM) at day 1
  Interventions: Biological: Ervebo
- Ervebo + Inmazeb (Experimental): Administration of Ervebo vaccine (72 million PFU IM) and Inmazeb IV (150 mg/kg) at day 1 and Inmazeb IV (150 mg/kg) at day 56
  Interventions: Biological: Ervebo; Biological: Inmazeb

INTERVENTIONS:
Biological: Ervebo — Ebola Zaire vaccine (rVSV∆G-ZEBOV-GP, live, attenuated) ≥ 72 million PFU, composed of the Indiana strain of recombinant vesicular stomatitis virus (rVSV) with a deletion of the envelope glycoprotein (G) of VSV replaced by the surface glycoprotein (GP) of the Kikwit 1995 strain of Ebola virus Zaire (ZEBOV)
  Other Names: r-VSV-ZEBOV vaccine
Biological: Inmazeb — Inmazeb (REGN-EB3), developed by Regeneron, is a cocktail of 3 neutralising humanised mAbs directed against 3 epitopes of the EBOV GP (atoltivimab, maftivimab and odesivimab). It is indicated for the treatment of EVD in adult patients (including pregnant women) and in children, including neonates born to mothers with confirmed EVD.
  Other Names: REGN-EB3
  Arms: Ervebo + Inmazeb

SUMMARY:
EBO-PEP is a multicentre, multi-epidemic, phase III, comparative, controlled, randomised, strict superiority trial in two unblinded parallel arms.

The trial will be open during EVD epidemics and will recruit asymptomatic participants at high risk of developing EVD.

Participants will be randomized (1:1) into one of two trial arms:

* Arm 1 (ERV): Ervebo D0 (72 million PFU IM)
* Arm 2 (ERV+IMZ): Ervebo D0 (72 million PFU IM) + Inmazeb IV (150 mg/kg) D0 + Ervebo D56 (revaccination)

Definition of high-risk:

Direct contact with a person with EBOV PCR-confirmed EVD with diarrhea, vomiting or external bleeding ("wet symptoms"), or with their body fluids; Direct contact with the dead body of a person with confirmed or probable EVD; Needlestick with a syringe contaminated by the blood of a person with confirmed or probable EVD; Or a child born to or breastfed by an individual with EVD

Trial follow-up All participants are monitored daily for a minimum of 21 days.

Some visits are conducted in person at the investigation site, also called the Post-Exposure Prophylaxis (PEP) center:

* at Day 5, Day 10, and Day 21 for the ERV arm,
* at Day 5, Day 10, Day 21, and Day 56 for the ERV+IMZ arm. Other visits are conducted at home or by phone, in collaboration with the Ministry of Health's surveillance team.

Participants in the ERV+IMZ arm have an in-person visit at Day 56 to be revaccinated with the Ervebo vaccine to compensate for potential inhibition of the vaccine response when Ervebo is administered simultaneously with Inmazeb.

Participants in the ERV arm have a phone visit at Day 56. For all participants, a phone visit is scheduled at Day 60. It corresponds to the last visit for all trial participants.

Follow-up in Case of Hospitalisation In case of clinical signs suggestive of EVD, participants enter the suspected case management pathway at the Ebola Treatment Center (ETC).

If EVD is confirmed by EBOV PCR, participants are allowed at the ETC, and their study samples are discontinued. They continue to be followed by the research team, and daily data are collected throughout their stay at the ETC until they are discharged alive or deceased. The day of discharge from the ETC marks the end of follow-up in the study for these participants.

Of note, participants in the ERV+IMZ arm who have confirmed EVD are not revaccinated at day 56.

Of note, participants in the ERV+IMZ arm who have confirmed EVD are not revaccinated at day 56.

If EVD is not confirmed, participants continue to be followed up by the PEP center according to the protocol.

DETAILED DESCRIPTION:
Since its discovery in the Democratic Republic of Congo (DRC) in 1976, the EBOV virus has been responsible for numerous epidemics. Outbreaks have occurred in the DRC, Gabon, Guinea, Liberia and Sierra Leone. Imported cases were also discovered in 1996 in South Africa, and in 2014 in Mali, Nigeria, Senegal, Italy, Spain, UK and USA (1). To date, the largest EVD epidemic occurred in West Africa between 2014 and 2016. It was responsible for over 28,000 infections and more than 11,000 deaths (2-4). Since this epidemic, EVD has emerged and re-emerged regularly in Sub-Saharan Africa (SSA).

Post-exposure prophylaxis (PEP) is the treatment of people at high risk of EVD. The main aim of PEP is to intervene during the asymptomatic incubation period (2-21 days) to prevent the development of EVD.

In addition to preventing the disease in individuals, an effective PEP strategy could reduce the rate of secondary attacks, thus interrupting transmission chains. If introduced rapidly, this tool could halt the spread of the disease and contribute to the fight against EVD epidemics (5). The particular vulnerability of healthcare personnel has been highlighted during several outbreaks, due to their close contact with infected patients and contaminated equipment (6). With an effective and accessible PEP tool, it will be possible to ensure the safety and protection of these essential personnel and minimize the risk of nosocomial transmission within healthcare establishments. PEP could also benefit contact tracing efforts by providing an appropriate preventive measure. By integrating PEP into comprehensive epidemic response strategies, it will be possible to improve countries' ability to control and mitigate the public health impact of EVD epidemics and prevent future outbreaks.

There is currently no comprehensive PEP strategy, i.e. one that combines several interventions. Several prophylactic interventions have been evaluated, including vaccination and mAb immunotherapy, each with its advantages and limitations (7-9). Although not intended for this use, Ervebo vaccine is currently administered as PEP during EVD epidemics, by being administered to contacts regardless of exposure levels.

MAbs have been administered as PEP on a compassionate basis, to healthcare workers following occupational exposure, in line with WHO expert advice from 2018 (10). In addition, mAbs are recommended as PEP for newborns of Ebola-infected mothers, within seven days of birth (11). PEP can prevent the risk of infection associated with a particular contact, but not the persistent risk of infection during an epidemic. A comprehensive strategy to protect high-risk contacts must therefore be put in place, including both a drug to prevent EVD after contact (mAb or antiviral) and a vaccine for long-term immunity, to guarantee both immediate and prolonged protection.

Inmazeb (REGN-EB3), developed by Regeneron, is a cocktail of 3 neutralizing humanized mAbs directed against 3 EBOV GP epitopes (atoltiviMab, maftiviMab and odesiviMab). It is indicated for the treatment of EVD in adult patients (including pregnant women) and in children, including neonates whose mothers have EVD at the time of delivery. Inmazeb inhibits viral entry into the target cell (12). This mechanism of action makes Inmazeb a promising candidate for PEP (34,40-44). In phase 1, the optimal dose was set at 150 mg/kg as a single intravenous (IV) dose, with good tolerability, except for moderate side effects such as headache and myalgia in 30% and 10% of participants respectively. The longest half-life of the three antibodies was 27.3 days (21.7 and 23.3 for the other two antibodies). At 180 days, the residual concentration of each antibody (administered at 150 mg/kg) is less than 10 mg/l (13). In the PALM trial, overall mortality after a single 150 mg/kg dose was estimated at 33.5% (versus 51.3% in the ZMapp control arm). However, the effect of treatment is strongly influenced by viral load. In patients with a high viral load at inclusion (NP Ct < 22), mortality was 63.6% (versus 86.2% in the Zmapp subgroup), while in patients with a low viral load at inclusion (NP Ct > 22), mortality was 11.2% (versus 25.8% in the Zmapp subgroup) (14). Following the PALM trial, Inmazeb was approved by the FDA for the treatment of EVD in adults and children (15).

A study conducted during the 10éme EVD epidemic in the DRC evaluated PEP with mAbs as part of a compassionate program (Post-Exposure Prophylaxis Monitored Emergency Used for Unregistered Intervention - PEP MEURI). In this study, 23 vaccine-naïve high-risk contacts received mAbs (21 Ebanga and 2 Inmazeb) after a median delay of one day between contact and PEP. At D14, none of the participants were symptom-free and their PCR was negative (16).

EBO-PEP is a multicentre, multi-epidemic, phase III, comparative, controlled, randomised, strict superiority trial in two unblinded parallel arms.

The trial will be open during EVD epidemics, and will recruit asymptomatic participants at high risk of developing EVD. Participants will be randomized (1:1) into one of two trial arms:

* Arm 1 (control arm): Ervebo D1 (72 million PFU IM)
* Arm 2: Ervebo D1 (72 million PFU IM) + Inmazeb IV (150 mg/kg) D1 + Ervebo D56 (revaccination)

Definition of high-risk:

Direct contact with a person with EBOV PCR-confirmed EVD with diarrhea, vomiting or external bleeding ("wet symptoms"), or with their body fluids; Direct contact with the dead body of a person with confirmed or probable EVD; Needlestick with a syringe contaminated by the blood of a person with confirmed or probable EVD; Or a child born to or breastfed by an individual with EVD

ELIGIBILITY:
Inclusion criteria

* Last high-risk contact within the last 5 days
* No sign or symptoms of EVD
* Signed and dated informed consent from participants over the age of majority to participate in the trial or from a representative of parental authority for minor participants.

Non-inclusion criteria

* History of vaccination with Ervebo or any other EVD vaccine within the last 5 years (self-reported by the participant)
* History of confirmed EVD within the last 5 years (self-reported by the participant)
* Hypersensitivity to any of the experimental medical products (IMP) or their excipients (self-reported by the participant)
* Participation in another therapeutic or vaccine trial for EVD
* Any other reason that, at the investigator's discretion, could compromise the participant's safety and cooperation in the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with EBOV PCR-confirmed symptomatic EVD | Between Day 1 and Day 21
  EVD rate

SECONDARY OUTCOMES:
Proportion of participants with EBOV PCR-confirmed symptomatic EVD | Between Day 1 and Day 60
  EVD rate
Safety and tolerance | Between Day 1 and Day 60
  Proportion of participants with a grade 3 or higher Adverse Event
Severity of EVD | Between Day 1 and Day 60
  Proportion of participants admitted to the Ebola Treatment Center with confirmed EVD meeting at least one of the following criteria:
  * Nucleoprotein cycle threshold (NP Ct) < 22
  * KDIGO stage 3
  * ASAT or ALAT > 5N
  * External bleeding
  * AVPU score
  * NEWS2 score ≥ 7
Proportion of participants with asymptomatic EVD | Between Day 1 and Day 21
  Rate of PCR-confirmed EVD
Proportion of deaths | Between Day 1 and Day 60
  Proportion of participants who died (all causes combined)
Changes in viral load | Between Day 1 and Day 21
  NP Ct curve (nucleoprotein cycle threshold)
Estimating cost-effectiveness | Between Day 1 and up to Day 60
  Incremental cost-effectiveness ratio (ICER) for ERV+IMZ arm vs ERV

CONTACTS AND LOCATIONS:
Overall Officials: Placide MBALA, MD, MSPH, PhD, Study Chair — INRB
Locations (4):
- National Institute for Biomedical Research (INRB), Kinshasa, Democratic Republic of the Congo
- Guinea Centre for Research and Training in Infectious Diseases (CERFIG), Conakry, Guinea
- National Public Health Institute of Liberia, Monrovia, Liberia
- University of Sierra Leone College of Medicine and Allied Health Sciences, Freetown, Sierra Leone

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huttner A, Agnandji ST, Combescure C, Fernandes JF, Bache EB, Kabwende L, Ndungu FM, Brosnahan J, Monath TP, Lemaitre B, Grillet S, Botto M, Engler O, Portmann J, Siegrist D, Bejon P, Silvera P, Kremsner P, Siegrist CA; VEBCON; VSV-EBOVAC; VSV-EBOPLUS Consortia. Determinants of antibody persistence across doses and continents after single-dose rVSV-ZEBOV vaccination for Ebola virus disease: an observational cohort study. Lancet Infect Dis. 2018 Jul;18(7):738-748. doi: 10.1016/S1473-3099(18)30165-8. Epub 2018 Apr 5. PMID 29627147
- [Background] Isa F, Gonzalez Ortiz AM, Meyer J, Hamilton JD, Olenchock BA, Brackin T, Ganguly S, Forleo-Neto E, Faria L, Heirman I, Marovich M, Hutter J, Polakowski L, Irvin SC, Thakur M, Hooper AT, Baum A, Petro CD, Fakih FA, McElrath MJ, De Rosa SC, Cohen KW, Williams LD, Hellman CA, Odeh AJ, Patel AH, Tomaras GD, Geba GP, Kyratsous CA, Musser B, Yancopoulos GD, Herman GA; Trial Working Group. Effect of timing of casirivimab and imdevimab administration relative to mRNA-1273 COVID-19 vaccination on vaccine-induced SARS-CoV-2 neutralising antibody responses: a prospective, open-label, phase 2, randomised controlled trial. Lancet Infect Dis. 2025 Jan;25(1):52-67. doi: 10.1016/S1473-3099(24)00421-3. Epub 2024 Sep 2. PMID 39236733
- [Background] Cao L, Li Y, Yang S, Li G, Zhou Q, Sun J, Xu T, Yang Y, Liao R, Shi Y, Yang Y, Zhu T, Huang S, Ji Y, Cong F, Luo Y, Zhu Y, Luan H, Zhang H, Chen J, Liu X, Luo R, Liu L, Wang P, Yu Y, Xing F, Ke B, Zheng H, Deng X, Zhang W, Lin C, Shi M, Li CM, Zhang Y, Zhang L, Dai J, Lu H, Zhao J, Zhang X, Guo D. The adenosine analog prodrug ATV006 is orally bioavailable and has preclinical efficacy against parental SARS-CoV-2 and variants. Sci Transl Med. 2022 Sep 7;14(661):eabm7621. doi: 10.1126/scitranslmed.abm7621. Epub 2022 Sep 7. PMID 35579533
- [Background] Jaspard M, Juchet S, Serra B, Mayoum B, Kanta IM, Camara MS, Mbala P, Kojan R, Malvy D. Post-exposure prophylaxis following high-risk contact with Ebola virus, using immunotherapies with monoclonal antibodies, in the eastern Democratic Republic of the Congo: an emergency use program. Int J Infect Dis. 2021 Dec;113:166-167. doi: 10.1016/j.ijid.2021.09.053. Epub 2021 Sep 26. PMID 34587535
- [Background] PREVAC Study Team; Kieh M, Richert L, Beavogui AH, Grund B, Leigh B, D'Ortenzio E, Doumbia S, Lhomme E, Sow S, Vatrinet R, Roy C, Kennedy SB, Faye S, Lees S, Millimouno NP, Camara AM, Samai M, Deen GF, Doumbia M, Esperou H, Pierson J, Watson-Jones D, Diallo A, Wentworth D, McLean C, Simon J, Wiedemann A, Dighero-Kemp B, Hensley L, Lane HC, Levy Y, Piot P, Greenwood B, Chene G, Neaton J, Yazdanpanah Y. Randomized Trial of Vaccines for Zaire Ebola Virus Disease. N Engl J Med. 2022 Dec 29;387(26):2411-2424. doi: 10.1056/NEJMoa2200072. Epub 2022 Dec 14. PMID 36516078
- [Background] Sivapalasingam S, Kamal M, Slim R, Hosain R, Shao W, Stoltz R, Yen J, Pologe LG, Cao Y, Partridge M, Sumner G, Lipsich L. Safety, pharmacokinetics, and immunogenicity of a co-formulated cocktail of three human monoclonal antibodies targeting Ebola virus glycoprotein in healthy adults: a randomised, first-in-human phase 1 study. Lancet Infect Dis. 2018 Aug;18(8):884-893. doi: 10.1016/S1473-3099(18)30397-9. Epub 2018 Jun 18. PMID 29929783
- [Background] Pascal KE, Dudgeon D, Trefry JC, Anantpadma M, Sakurai Y, Murin CD, Turner HL, Fairhurst J, Torres M, Rafique A, Yan Y, Badithe A, Yu K, Potocky T, Bixler SL, Chance TB, Pratt WD, Rossi FD, Shamblin JD, Wollen SE, Zelko JM, Carrion R Jr, Worwa G, Staples HM, Burakov D, Babb R, Chen G, Martin J, Huang TT, Erlandson K, Willis MS, Armstrong K, Dreier TM, Ward AB, Davey RA, Pitt MLM, Lipsich L, Mason P, Olson W, Stahl N, Kyratsous CA. Development of Clinical-Stage Human Monoclonal Antibodies That Treat Advanced Ebola Virus Disease in Nonhuman Primates. J Infect Dis. 2018 Nov 22;218(suppl_5):S612-S626. doi: 10.1093/infdis/jiy285. PMID 29860496
- [Background] Moso MA, Lim CK, Williams E, Marshall C, McCarthy J, Williamson DA. Prevention and post-exposure management of occupational exposure to Ebola virus. Lancet Infect Dis. 2024 Feb;24(2):e93-e105. doi: 10.1016/S1473-3099(23)00376-6. Epub 2023 Sep 15. PMID 37722397
- [Background] Crozier I, Britson KA, Wolfe DN, Klena JD, Hensley LE, Lee JS, Wolfraim LA, Taylor KL, Higgs ES, Montgomery JM, Martins KA. The Evolution of Medical Countermeasures for Ebola Virus Disease: Lessons Learned and Next Steps. Vaccines (Basel). 2022 Jul 29;10(8):1213. doi: 10.3390/vaccines10081213. PMID 36016101
- [Background] Fischer WA 2nd, Vetter P, Bausch DG, Burgess T, Davey RT Jr, Fowler R, Hayden FG, Jahrling PB, Kalil AC, Mayers DL, Mehta AK, Uyeki TM, Jacobs M. Ebola virus disease: an update on post-exposure prophylaxis. Lancet Infect Dis. 2018 Jun;18(6):e183-e192. doi: 10.1016/S1473-3099(17)30677-1. Epub 2017 Nov 15. PMID 29153266
- [Background] Bower H, Johnson S, Bangura MS, Kamara AJ, Kamara O, Mansaray SH, Sesay D, Turay C, Checchi F, Glynn JR. Exposure-Specific and Age-Specific Attack Rates for Ebola Virus Disease in Ebola-Affected Households, Sierra Leone. Emerg Infect Dis. 2016 Aug;22(8):1403-11. doi: 10.3201/eid2208.160163. Epub 2016 Aug 15. PMID 27144428
- [Background] Hoffmann Dahl E, Mbala P, Juchet S, Toure A, Montoyo A, Serra B, Kojan R, D'Ortenzio E, Blomberg B, Jaspard M. Improving Ebola virus disease outbreak control through targeted post-exposure prophylaxis. Lancet Glob Health. 2024 Oct;12(10):e1730-e1736. doi: 10.1016/S2214-109X(24)00255-9. Epub 2024 Sep 10. PMID 39270687
- [Background] Languon S, Quaye O. Filovirus Disease Outbreaks: A Chronological Overview. Virology (Auckl). 2019 Jun 21;10:1178122X19849927. doi: 10.1177/1178122X19849927. eCollection 2019. PMID 31258326
- See also: 2.WHO | Regional Office for Africa [Internet]. 2024 [cited 30 juill 2024]. Ebola Disease — https://www.afro.who.int/health-topics/ebola-disease
- See also: 3.CDC. Ebola. 2024 [cited 4 oct 2024]. Outbreak History. — https://www.cdc.gov/ebola/outbreaks/index.html
- See also: 11. Therapeutics for Ebola virus disease [Internet]. [cited 4 oct 2024] — https://www.who.int/publications/i/item/9789240055742
- See also: 22. Implementation and management of contact tracing for Ebola virus disease [Internet]. [cited 4 oct 2024]. — https://www.who.int/publications/i/item/WHO-EVD-Guidance-Contact-15.1
- See also: 25. Study Details | Pilot Study Evaluating the Impact of Delay Between Administration of Inmazeb Administration and Vaccination by Ervebo on Vaccine Immune Response on Healthy Volunteers | ClinicalTrials.gov — https://clinicaltrials.gov/study/NCT05202288?term=NCT05202288&rank=1